CLINICAL TRIAL: NCT05841004
Title: A Randomized, Crossover Study Confirming Performance of a New Single-use Compact Intermittent Catheter vs. Infyna Chic in a Pop-ulation of Adult Female Intermittent Catheter Users.
Brief Title: Clinical Trial of New Single-use Compact Intermittent Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CP356
Record Dates: First submitted 2023-03-24; First posted 2023-05-03 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-12

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: controlled crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational device - newly developed intermittent compact catheter (Experimental): Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (CH12 and CH14) for urinary drainage. The investigational device is for single use.
  Interventions: Device: Investigational device; Device: Comparator device
- Hollister Infyna Chic (Active Comparator): The comparator is Hollister Infyna Chic, a CE-marked single-use compact catheter.
  Interventions: Device: Investigational device; Device: Comparator device

INTERVENTIONS:
Device: Investigational device — Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The investigational device is for single use.
Device: Comparator device — Hollister Infyna Chic, single-use compact catheter.

SUMMARY:
The study is a randomised, single-blinded, controlled crossover study. The total study duration for the individual subject will be between two days - two weeks, consisting of three site visits. Visits 0 and 1 can be performed on the same day. Visit 2 can be performed the day after visit 1. For visit 1 and 2, catheterizations will be performed in a hospital setting by a health care professional for bladder emptying assessment and collection of urine samples for haematuria assessment. A sub-group of subjects (all enrolled subjects at DK sites) will be asked to conduct a self-catheterization at visit 2 after hcp catheterization and evaluate discomfort and PVR.

The total study duration for the individual subject will be up to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Is Female
* Is at least 18 years of age and has full legal capacity
* Has signed an informed consent form
* Has used clean intermittent self-catheterisation (CISC) (CH12 or CH14) for at least one month up to inclusion
* Is using intermittent self-catheterisation for a minimum of 3 times per day for bladder emptying
* Has used a compact catheter 50% of the time (or more) for the last two weeks prior to entering the study
* Has the ability (assessed by investigator) and willingness to follow study procedures or is able to use a compact catheter assessed by investigator

Exclusion Criteria:

* Is participating in any other clinical study during this investigation
* Has previously participated in this study
* Has symptoms of urinary tract infection at time of inclusion, as judged by the investigator (if the patient recovers within the recruitment period, a second inclusion is allowed, under a different subject id)
* Is an individual with a history of - suspected to be - or showing signs of producing an excessive amount of mucus or large/clustered sediments or debris
* Has any known allergies towards ingredients in the investigational device
* Is pregnant
* Is breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karin Andersen, MD, Principal Investigator — Odense Universitetshospital
Locations (1):
- Odense Universitetshospital, Odense, Denmark

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational Device First, Then Hollister Infyna Chic: Investigational device: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The investigational device is for single use.
  Comparator device: Hollister Infyna Chic, single-use compact catheter.
- Hollister Infyna Chic, Then Investigational Device: The comparator is Hollister Infyna Chic, a CE-marked single-use compact catheter.
  Comparator device: Hollister Infyna Chic, single-use compact catheter.
  Investigational device: Ready-to-use, sterile, hydrophilic coated intermittent female compact catheter (sizes CH12 and CH14) for urinary drainage. The investigational device is for single use.
Period: First Intervention (Visit 1)
Arm/Group | Investigational Device First, Then Hollister Infyna Chic | Hollister Infyna Chic, Then Investigational Device
Started | 37 | 36
Completed | 36 | 36
Not Completed | 1 | 0
Period: Second Intervention (Visit 2)
Arm/Group | Investigational Device First, Then Hollister Infyna Chic | Hollister Infyna Chic, Then Investigational Device
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total ITT Population Baseline Measures: As this study was a crossover study, each participant underwent catheterizations with both the investigational device and the comparator device. The study consisted of three study visits (V0-V2) . Visit 0 included subject enrollment, and randomization. Randomization was done centralized, randomly assigning subjects to two intervention sequences. Hence, the first group used the investigational device at the first follow-up visit (V1). Subsequently, the comparator device was used at the visit 2 which also terminated the study. The second group tested the devices in reversed order. The total study duration was up to two weeks for the individual subject
Arm/Group | Total ITT Population Baseline Measures
Number analyzed (Participants) | 73
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 57
  United Kingdom | 16

OUTCOME MEASURES:

1. Primary Outcome: Residual Volume at 1st Flow-stop (Catheterisation Performed by HCP)
Description: Measure residual volume at 1st flow-stop i.e., post catheterisation volume minus volume at 1st flow-stop, both derived from a catheterisation profile, [mL]
Time Frame: At Visit 1 and Visit 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mL
Arm/Group | Investigational Device - Newly Developed Intermittent Compact Catheter | Hollister Infyna Chic
Number analyzed (Participants) | 72 | 72
mL | 15.3 [3.7 to 26.9] | 23.7 [10.8 to 37.0]

2. Secondary Outcome: Number of Flowstops (Catheterisation Performed by a Healthcare Professional)
Description: Measure number of flow-stop episodes derived from a catheterisation profile (catheterisation performed by a healthcare professional), [number].
Time Frame: At Visit 1 and Visit 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of flow-stops
Arm/Group | Investigational Device - Newly Developed Intermittent Compact Catheter | Hollister Infyna Chic
Number analyzed (Participants) | 72 | 72
Number of flow-stops | 0.27 [0.13 to 0.55] | 0.59 [0.36 to 0.96]

3. Secondary Outcome: Residual Volume Post Catheterisation
Description: Measure average residual volume post catheterisation (PVR) measured with a bladder scanner (triplicate measurements), [mL],
Time Frame: At Visit 1 and Visit 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Investigational Device - Newly Developed Intermittent Compact Catheter | Hollister Infyna Chic
Number analyzed (Participants) | 72 | 72
mL | 10.1 (34.1) | 15.8 (51.0)

4. Secondary Outcome: Number of Adverse Events
Description: Count number of Adverse events, [number]
Time Frame: At Visit 1 and Visit 2
Measure: Number; unit: Adverse events
Arm/Group | Investigational Device - Newly Developed Intermittent Compact Catheter | Hollister Infyna Chic
Number analyzed (Participants) | 72 | 72
Adverse events | 1 | 1

5. Other Pre Specified Outcome: Discomfort Measure by VAS (Only in DK)
Description: Discomfort is measured by Visual Analogue Scale (VAS), which is measured on a 10 cm horizontal scale ranging from "no discomfort" at 0 cm to "worst possible discomfort" at 10 cm caused by the catheter, by drawing a vertical line indicating how the subject experienced the catheterization divided into the four following categories: Discomfort at insertion measured using the VAS (VAS) [cm] Discomfort at withdrawal measured using the VAS, [cm] Discomfort during emptying of bladder measured using the VAS, [cm] Discomfort at end of emptying the bladder measured using the VAS, [cm]
Time Frame: At Visit 1 and Visit 2
Population: This analysis was only performed with the investigational device and only on the participants from sites in Denmark.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigational Device - Newly Developed Intermittent Compact Catheter | Hollister Infyna Chic
Number analyzed (Participants) | 54 | 0
score on a scale
  Discomfort at insertion | 0.19 (0.51) |
  Discomfort at withdrawal | 0.24 (1.02) |
  Discomfort by completion | 0.21 (0.62) |
  Discomfort when emptying | 0.19 (0.76) |

6. Post Hoc Outcome: Response to Treatment, Residual Volume of Urine at First Flow-stop Under 10 Milliliter
Description: Responder analysis involved testing the proportion of all catheterisations which achieved a residual volume of urine at first flow-stop of less than 10 milliliter.
  In this clinical investigation, responder analyses were introduced as an expansion of the data analyses due to the few extreme RV1 values, which presented a challenge to the predetermined statistical model. (see 'limitations and caveats' section for further details). Responder analyses evaluated the proportion of patients who achieved the positive treatment response threshold, highlighting individual patient responses rather than average effects across the entire population. Successful treatment responses were defined as individuals who achieved the desired outcome of catheterisation, i.e., complete and effective bladder emptying without repositioning, in terms flow-stops defined as zero flow-stops and in terms of complete emptying of the bladder was defined as an RV1<10 mL.
Time Frame: At Visit 1 and Visit 2
Measure: Mean (95% Confidence Interval); unit: percentage of catheterisations
Arm/Group | Investigational Device - Newly Developed Intermittent Compact Catheter | Hollister Infyna Chic
Number analyzed (Participants) | 72 | 72
percentage of catheterisations | 84 [72 to 91] | 68 [56 to 79]

7. Post Hoc Outcome: Response to Treatment, 0 Flow-stops
Description: Responder analysis involved testing the proportion of all catheterisations which did not experience any flow-stops.
  In this clinical investigation, responder analyses were introduced as an expansion of the data analyses due to the few extreme RV1 values, which presented a challenge to the predetermined statistical model. (see 'limitations and caveats' section for further details). Responder analyses evaluated the proportion of patients who achieved the positive treatment response threshold, highlighting individual patient responses rather than average effects across the entire population. Successful treatment responses were defined as individuals who achieved the desired outcome of catheterisation, i.e., complete and effective bladder emptying without repositioning, in terms flow-stops defined as zero flow-stops and in terms of complete emptying of the bladder was defined as an RV1<10 mL.
Time Frame: At Visit 1 and Visit 2
Measure: Mean (95% Confidence Interval); unit: percentage of catheterisations
Arm/Group | Investigational Device - Newly Developed Intermittent Compact Catheter | Hollister Infyna Chic
Number analyzed (Participants) | 72 | 72
percentage of catheterisations | 87 [76 to 93] | 61 [48 to 72]

ADVERSE EVENTS:
Time Frame: Adverse events were registered from the individual's enrolment until termination in the study. The total study duration for the individual subject was between two days to two weeks, consisting of three site visits (V0-V2).
Arm/Group | Investigational Device - Newly Developed Intermittent Compact Catheter | Hollister Infyna Chic
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/72
Other Adverse Events (participants affected / at risk) | 1/73 | 1/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device - Newly Developed Intermittent Compact Catheter (N=73) | Hollister Infyna Chic (N=72)
Obstipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain when urinating (Renal and urinary disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The natural distribution of residual volume at 1st flow-stop values skews positively. This carries a high risk of influence by random occurrences of extreme values. These can occur without systematic relation to product or subject and can obscure interpretability of the analysis. To counter this effect, post hoc responder analyses were included, testing the benefit of treatment through the proportion of individuals who achieve the desired outcome, i.e., complete and effective bladder drainage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/04/NCT05841004/Prot_SAP_000.pdf